CLINICAL TRIAL: NCT01297998
Title: A Phase I Study of Adjuvant Chemotherapy With Gemcitabine Plus Cisplatin in Patients With Biliary Tract Cancer Undergoing Curative Resection Without Major Hepatectomy
Brief Title: A Phase I Study of Adjuvant Chemotherapy With GC in Biliary Tract Cancer Undergoing Resection Without Major Hepatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1004; UMIN000004622 (Registry Identifier: UMIN)
Record Dates: First submitted 2011-02-07; First posted 2011-02-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2014-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine , cisplatin (Experimental)
  Interventions: Drug: gemcitabine , cisplatin

INTERVENTIONS:
Drug: gemcitabine , cisplatin — Dose of gemcitabine and cisplatin and treatment schedule
  Other Names: Gemcitabine;gemzer,Cisplatin;Cispulan

SUMMARY:
To decide maximum tolerated dose and recommended dose of treatment using gemcitabine plus cisplatin combination therapy in patients with biliary tract cancer undergoing resection without major hepatectomy.

DETAILED DESCRIPTION:
Surgery currently remains the only potentially curative treatment for biliary tract cancer (BTC), and most patients develop recurrence. Therefore, effective adjuvant chemotherapy is required to increase the curability of surgery and to prolong the survival in these patients. However, to date, no standard adjuvant chemotherapy has been established, and a guideline for BTC treatment recommends that trials of adjuvant chemotherapy be carried out.

Based on results from clinical studies in unresectable BTC, gemcitabine, platinum agent, fluoropyrimidine are considered to have activity against BTC. These agents are expected to be effective in the postoperative adjuvant therapy for BTC, Thus, randomized controlled trials with gemcitabine are ongoing, and the results are expected. Recently, in the ABC-02 study, the first prospective multicenter phase III study in patients with unresectable BTC, gemcitabine/cisplatin combination chemotherapy was compared with gemcitabine monotherapy and showed that the combination therapy significantly prolonged MST (from 8.1 to 11.7 months; P < 0.001). Gemcitabine/cisplatin combination therapy is now considered to be the standard regimen for unresectable BTC, and we expect this regimen to be effective for postoperative adjuvant therapy.

Though hepatectomy is frequently performed in surgery for BTC, it is unclear that the effect of anticancer agent is affected by hepatectomy. Because gemcitabine is metabolized by cytidine deaminase primarily in the liver, it considered to have decreased the metabolic ability of gemcitabine after hepatectomy. Some clinical studies demonstrated that patient with hepatectomy could not tolerate the standard dose and schedule of gemcitabine. In the adjuvant chemotherapy with gemcitabine, it is necessary to examine separately whether hepatectomy was undergone or not.

In this study, we aimed to assess the safety and efficacy of gemcitabine/cisplatin combination chemotherapy in patients with biliary tract cancer undergoing curative resection without hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Biliary tract cancer (BTC) with more than stage IB
2. BTC undergoing R0 or R1 resection without major hepatectomy
3. Older than 20 years old
4. PS0 or 1
5. No treatment other than surgery
6. No dysfunction of main organs
7. Possible oral intake
8. Treatment start; after 4 weeks and within 12 weeks after surgery
9. Obtained written informed consent

Exclusion Criteria:

1. Patients with resection of major hepatectomy
2. Patients with double cancers
3. Patients having severe allergy
4. Patients with severe organ dysfunction
5. Patients with active infectious disease
6. Pregnancy
7. Patients with severe psychological disease
8. Patients seem inadequate for this study by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Within 2 courses (every 2 weeks in Level -2 and -1; every 3 weeks in Level 0 and 1)
  To establish the maximum tolerated dose of gemcitabine plus cisplatin in patients with biliary tract cancer undergoing curative resection without major hepatectomy

SECONDARY OUTCOMES:
Number of Participants with dose limiting toxicity | At the end of adjuvant chemotherapy (6 months)
  Dose limiting toxicity is defined as follows
  1. Grade 4 neutropenia, thrombocytopenia
  2. Grade 3 or 4 febrile neutropenia
  3. Grade 3 or 4 non-hematological adverse events unless unresponsive to treatment
  4. Any adverse events resulting in interruption of dosing on day 8 in both the two courses
  5. Any adverse events resulting in dose modification or delay of longer than 2 week

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuo Ajiki, MD, PhD, Study Director — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Kobe, Japan

REFERENCES:
- [Derived] Toyoda M, Ajiki T, Fujiwara Y, Nagano H, Kobayashi S, Sakai D, Hatano E, Kanai M, Nakamori S, Miyamoto A, Tsuji A, Kaihara S, Ikoma H, Takemura S, Toyokawa H, Terajima H, Morita S, Ioka T. Phase I study of adjuvant chemotherapy with gemcitabine plus cisplatin in patients with biliary tract cancer undergoing curative resection without major hepatectomy (KHBO1004). Cancer Chemother Pharmacol. 2014 Jun;73(6):1295-301. doi: 10.1007/s00280-014-2431-y. Epub 2014 Mar 11. PMID 24614947